CLINICAL TRIAL: NCT07056998
Title: Accuracy of Artificial Intelligence Technology in Detecting the Quality of Endodontic Treatment Diagnostic Accuracy Experimental Study.
Brief Title: On Previously Root Canal-treated Patients Using an AI Program, Detect the Accuracy of it in the Detection of Root Canal Obturation Quality on CBCT Compared With Conventional PA Radiography, e.g., Voids, Length of Obturation, and Density, and Then do Retreatment if Any Failure is Recorded.
Acronym: AI
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Tala Ghassan Hassan Odeh (Other)
Responsible Party: Sponsor-Investigator, Tala Ghassan Hassan Odeh, B.D.S. Dental College, Future University in Egypt
Organization: Future University in Egypt (Other)
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Diagnostic
Other Study IDs: FUE.REC(44)/11-2024
Record Dates: First submitted 2025-06-25; First posted 2025-07-09 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Root Canal Treatment
Keywords: quality of root canal , Artificial intelligence, CBCT

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Length of Root Filling (Active Comparator): 1. Length of Root Filling Ideal: 0-2 mm short of the radiographic apex Overfilling: Beyond the apex - may lead to periapical irritation Underfilling: More than 2 mm short - associated with poor prognosis Measuring unit: millimeters (mm) from the radiographic apex
  Interventions: Procedure: root canal retreatment
- Density/Homogeneity (Active Comparator): Criteria: No visible voids in: Canal system, Between gutta-percha and canal wall Assessment: Radiographic inspection (digital or analog) Measuring tool: Qualitative (visual rating) or CBCT grayscale values for homogeneity
  Interventions: Procedure: root canal retreatment
- Presence of Voids (Active Comparator): Criteria: Voids indicate poor condensation or adaptation Assessment tools: Periapical radiographs, CBCT. Measuring unit: Number, size (mm or μm), or volume (%) of voids
  Interventions: Procedure: root canal retreatment

INTERVENTIONS:
Procedure: root canal retreatment — if Retreatment was needed, local anesthesia using 1.8 ml (one cartridge) of 4% articaine with 1:100,000 epinephrine local anesthetic solution, administered with end -loading cartridge aspirating syringe and a 27-gauge long needle. Under rubber dam isolation, All carious tissue and existing coronal restorations were thoroughly removed using a round bur, an endodontic access cavity, canal preparation and removal of existing root canal filling, irrigation with 2.6% NAOCL and saline, determining the working length using apex locator and PA radiograph, to be 0.5 to 1 mm shorter than radiographic apex, Drying the canal with paper point and obturation to achieve a dense, well adapted Monoblock obturation. A post-obturation periapical radiograph was taken to confirm the quality of the fill in terms of length, density, then sealed by a temporary restorative material.

SUMMARY:
aims to evaluate the accuracy of clinicians (conventional radiograph) compared to cone beam computed tomography (CBCT) and artificial intelligence software's ability to identify the quality of root canal obturation. Will the use of artificial intelligence software be compared to conventional software in accuracy?

DETAILED DESCRIPTION:
AI is a new method used in the medical field, specifically dentistry. aiming to detect the accuracy of AI in the field of endodontics, specifically in root canal quality (correct length, density, taper, and coronal seal) compared to the skill of the endodontist using 2D radiograph and CBCT, and if any signs and symptoms of failure are detected in the treatment, retreatment is done according to the needs of each case.

ELIGIBILITY:
Inclusion Criteria:

1. Medically free patients with no systemic disease: (American Society of Anesthesiologists / (ASA Class I or II).
2. Age range is between18 to 50 years
3. No sex predilection.
4. All patients must have good oral hygiene. 5 -patients with root canal-treated teeth.

6- restorable teeth. 7- Positive patient acceptance for participating in the study. 8- Patients can sign informed consent.

Exclusion Criteria:

* 1-Patients with very poor oral hygiene. 2-Patients above 50 years and below 18 years. 3-Pregnant and lactating women 4-Psychologically disturbed patients. 5-nonrestorable teeth.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 3 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
root canal quality Length of Root Filling | preprocedural(day 1) and if treatment needed after the completion of the it up to 1month
  Length of Root Filling Ideal: 0-2 mm short of the radiographic apex Overfilling: Beyond the apex - may lead to periapical irritation Underfilling: More than 2 mm short - associated with poor prognosis Measuring unit: millimeters (mm) from the radiographic apex

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Oral and Dental Medicine future university, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
only IPD used in the results publication
Supporting Information: Study Protocol, ICF
Time Frame: Beginning of 2026, a year after publication, with no end date